CLINICAL TRIAL: NCT01297140
Title: The Role of Personality in the Occurrence of Behavioural Disorders in Patients Suffering From Alzheimer Disease
Brief Title: The PACO Study ("Personnalité Alzheimer COmportement")
Acronym: PACO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2008.508
Record Dates: First submitted 2011-02-14; First posted 2011-02-16 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-10

CONDITIONS: Alzheimer Disease
Keywords: Psychiatry; Behaviour; Alzheimer's; Personality
MeSH Terms: conditions — Alzheimer Disease; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- questionary (Experimental)
  Interventions: Behavioral: questioning

INTERVENTIONS:
Behavioral: questioning — Patients will be screened by questioning them and their caregiver and from the results of the clinical examination and the biological and neuroradiological tests habitually carried out in cases of dementia and following accepted procedures.

SUMMARY:
Alzheimer's disease is characterised by a loss of cognitive functions and behavioural problems as set out under the term "Behavioural and psychological symptoms of dementia (BPSD)". The impact of BPSD in everyday life has heavy consequences for the patient and their family. The precocity of incidence, the frequency and the intensity of the BPSD are associated with a rapid decline in cognitive functions, an alteration in the activities of daily living, and a decrease in the quality of life for both the patient and the helper, an increased risk of hospitalisation and of institutionalisation as well as an increase in the cost to the health system. A greater understanding of the risk factors for the occurence of the BPSD would better allow the detection of patients who are particularly at risk for BPSD, to anticipate the crisis situations by proposing early and adapted care, and to better target the medicinal therapies. Certain observational arguments or results of retrospective studies speak in favour of the role of the basic personality in the occurence of BPSD in Alzheimer's disease. The investigators propose to clarify this role through a prospective study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged over 50 years ;
* In-patient or out-patient at one of the centres participating in the study ;
* Meeting all the diagnostic criteria for dementia due to AD (NINCDS ADRDA, CDR 1 or 2) or pre-dementia with a CDR of 0.5 (Berr et al., 2006, Dubois et al, 2007) ;
* Covered by the state's Social Security system ;
* With sufficient visual, auditory and oral and written French language skills to complete the clinical and neuropsychological evaluations ;
* Accompanied by a caregiver in sufficient contact with the subject to be able to assess their personality and note the onset of changes in behaviour.

Exclusion Criteria:

* Patients with a progressive and/or poorly managed psychiatric pathology (patients with stabilised depression could be included in the study) ;
* Patients taking any neuroleptic psychotropic medication ;
* Patients taking other psychotropic medication, with the exception of any antidepressant, hypnotic, anxiolytic, acetylcholinesterase inhibitors or Memantine which has been prescribed and stabilised for more than 3 months
* Patients with forms of dementia with an aetiology other than that of Alzheimer's disease (frontotemporal dementia, vascular dementia, Lewy Body dementia, and types of dementia that arise as a result of an underlying untreated disease, such as dysthyroidism, vitamin B12 or folic acid deficiency, syphilis, anaemia or hydroelectrolytic disorders) ;
* Patients with serious, progressive or unstable pathologies which could interfere with the variables under consideration ;
* Deafness or blindness which could compromise evaluation of the patient ;
* Pregnancy ;
* Patients under any type of guardianship or belonging to a restricted category as laid out in the Public Health Code ;
* Patients without a suitable caregiver willing to participate.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2009-01; Primary Completion 2015-07 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Behavioural and psychological symptoms of dementia (BPSD) | 18 months
  To measure (at inclusion, and at 6, 12, 18 months) the effect of premorbid personality and life events on the likelihood of a patient with probable Alzheimer's disease being affected by each of the BPSD categories: hyperactivity, psychotic symptoms, mood symptoms and apathy.

SECONDARY OUTCOMES:
social cognition tests | during the inclusion visit
  To evaluate, at the time of inclusion, the connection between the basic personality and the performance in social cognition tests (capacity to interact with others)
connection between social cognitive tests and BPSD | 18 months
  To evaluate (at inclusion and after 6, 12, 18 months) the connection between the performance of the social cognitive tests at the time of inclusion and the risks of occurrence of BPSD.
connection between cerebral atrophy and BPSD | 18 months
  To evaluate the connection between the distribution of regional cerebral atrophy, determined by a MRI at the time of inclusion, and the risk of subsequent BPSD.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Gériatrie - Hôpital des Charpennes - Hospices Civils de Lyon, Villeurbanne, France

REFERENCES:
- [Derived] Rouch I, Dorey JM, Boublay N, Henaff MA, Dibie-Racoupeau F, Makaroff Z, Harston S, Benoit M, Barrellon MO, Federico D, Laurent B, Padovan C, Krolak-Salmon P; PACO group. Personality, Alzheimer's disease and behavioural and cognitive symptoms of dementia: the PACO prospective cohort study protocol. BMC Geriatr. 2014 Oct 10;14:110. doi: 10.1186/1471-2318-14-110. PMID 25304446